CLINICAL TRIAL: NCT04693819
Title: Exploratory Study on the Role of Somatic Modulation in Hyperacusis
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: SomHyp
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2020-12

CONDITIONS: Hyperacusis
Keywords: Hyperacusis; Somatic; Modulation
MeSH Terms: conditions — Hyperacusis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperacusis: Abnormally reduced tolerance to sound
  Interventions: Diagnostic Test: Somatic modulation

INTERVENTIONS:
Diagnostic Test: Somatic modulation — Type of modulations: 3 jaw and 6 cervical spine modulations, 1 control movement (i.e. without any expected somatic modulation effect) Jaw modulations: laterotrusion to the left, laterotrusion to the right and protrusion Cervical spine modulations: isometric flexion, extension and left and right lateroflexion of the head against resistance of the investigator's hand, compression and traction of the cervical spine in sitting position.
  Control movement: the investigator's hand rests against the patient's forehead without any force application

SUMMARY:
This study focuses on patients with a primary complaint of hyperacusis. Hyperacusis has been defined as 'abnormally reduced tolerance to sound' and is commonly associated with tinnitus. The effects of somatic modulation upon tinnitus have been studied, but not so for hyperacusis.. The effect of 9 somatic modulations (i.e. 3 jaw modulations and 6 cervical spine modulations) and 1 control movement (i.e. without any somatic modulation effect) in random order on the sound tolerance of a 1 kilohertz (kHz) broadband noise sound and the tinnitus experience will be investigated. More specifically, the perceived loudness and intrusiveness of this sound and the tinnitus sound will be evaluated before somatic modulation and during the somatic modulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of hyperacusis

Exclusion Criteria:

* Primary complaint of tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be aimed at adults experiencing a primary complaint of hyperacusis (i.e. abnormally reduced tolerance to sound).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in rating of hyperacusis (loudness and intrusiveness) after modulation | Baseline (Before modulation), Immediately after modulation
  Change in hyperacusis loudness and intrusiveness rating by use of a visual analogue scale

SECONDARY OUTCOMES:
Change in rating of tinnitus (loudness and intrusiveness) after modulation | Baseline (Before modulation), Immediately after modulation
  Change in tinnitus loudness and intrusiveness rating by use of a visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shore SE. Plasticity of somatosensory inputs to the cochlear nucleus--implications for tinnitus. Hear Res. 2011 Nov;281(1-2):38-46. doi: 10.1016/j.heares.2011.05.001. Epub 2011 May 18. PMID 21620940
- [Background] Baguley DM, Hoare DJ. Hyperacusis: major research questions. HNO. 2018 May;66(5):358-363. doi: 10.1007/s00106-017-0464-3. PMID 29392341
- [Background] Baguley DM. Hyperacusis. J R Soc Med. 2003 Dec;96(12):582-5. doi: 10.1177/014107680309601203. No abstract available. PMID 14645606
- [Derived] Demoen S, Michiels S, Gilles A, Vermeersch H, Joossen I, Vanderveken OM, Lammers MJW, Timmermans A, Van Rompaey V, Baguley D, Jacquemin L. Pilot study on the role of somatic modulation in hyperacusis. Eur Arch Otorhinolaryngol. 2023 Mar;280(3):1425-1435. doi: 10.1007/s00405-022-07695-y. Epub 2022 Oct 13. PMID 36224398